CLINICAL TRIAL: NCT04752098
Title: Assessment of Metabolic Bone Disease of Prematurity Using an Acoustic Method
Brief Title: A Study to Assess Metabolic Bone Disease of Prematurity Using an Acoustic Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Azra Alizad, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-001498; 1R21AR075370-01A1 (NIH); 5R21AR075370-02 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Bone Disease; Osteopenia; Neonatal Rickets
Keywords: Bone Diseases; bone health; Fracture; infancy; Low Birth Weight Infant; mineralization; Neonatal; Pediatrics; Premature; ultrasound; Rickets
MeSH Terms: conditions — Bone Diseases, Metabolic; Bone Diseases; Fractures, Bone; Calcinosis; Premature Birth; Rickets | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Children (Newborns born full term (males and females), and infants born preterm (males and females)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- premature infants and full term infants (Other): The study visits will be at ≥3 time points at ages: within the first 28 days after birth, 2 months, 3 months, and, if still hospitalized, at 4 months and at 6 months.
  * The ultrasound machine to the nursery or neonatal intensive care unit at a scheduled time.
  * The appropriate ultrasound probe will be placed on the infant's tibia and a miniature hydrophone near the probe. A series of ultrasound measurements will be obtained and the ultrasound data will be saved for offline processing.
  * The Investigators will repeat the measurement in 3 locations of the infant's tibia.
  * Each ultrasound measurement takes a few seconds. The complete ultrasound study will take about 15 minutes at each visit.
  * All procedures will be conducted in the nursery or neonatal intensive care unit to ensure infant safety.
  * The ultrasound measurement for full-term infants can be done in ultrasound lab.
  Interventions: Diagnostic Test: Vibro-acoustic analysis (VAA), based on ultrasound radiation force

INTERVENTIONS:
Diagnostic Test: Vibro-acoustic analysis (VAA), based on ultrasound radiation force — The study will develop and validate a new ultrasonic method for assessment of infant bone by evaluating structural and mechanical characteristics of the infant tibia. This project will utilize a novel, non-invasive method, vibro-acoustic analysis (VAA), to evaluate infant bone properties in a wide frequency range while reducing the artifacts from soft tissue.
  Other Names: ultrasound

SUMMARY:
The goal of this project is to develop a new noninvasive ultrasound based technique, called vibro-acoustic analysis (VAA), for evaluation of infant bone health with particular application in assessment of bone health in premature infants who are at risk for bone disease.

DETAILED DESCRIPTION:
With increased survival of very low birth weight and premature infants over recent decades, bone assessment has become especially vital with the recognition of metabolic bone disease (MBD) of prematurity. Bone assessment became especially vital during last decades with the growing emphasis on metabolic bone disease of prematurity and low-birth-weight infants. Statistics shows that up to 50% of low birth weight and preterm newborns are likely to develop metabolic bone disease. Currently, no screening test has been shown to provide both sensitive and specific evidence of developing MBD over the first several weeks of life in the premature infants. Therefore, there is a need for a non-invasive tool for evaluation of infant bone health. This study will be conducted on premature infants at risk for MBD at multiple time points during their growth, with full term infants as controls. vibro-acoustic analysis (VAA) measurements will be done on the tibia. VAA measurements for the premature infants will be compared to those of full term infants. Performance of VAA in identifying osteopenia and its ability to monitor the response to treatment will be evaluated. The investigators will use an ultrasound system that has been used in the pilot study and employ a transducer with a smaller footprint for pediatric application.

ELIGIBILITY:
Inclusion Criteria:

* Full term newborns, approximately equal number of male and female newborn, age <28 days.
* Preterm infants, approximately equal number of male and female preterm infants with gestational age at birth <37 weeks or birth weight <1500 grams.

Exclusion Criteria:

* Infants currently requiring continuous cardiovascular medication infusions, including but not limited to, dopamine, epinephrine, milrinone, and dobutamine (may have received these medications in the past.
* Infants with major congenital anomalies that may affect bone health or structure.
* For full term infants, infants with a history of intrauterine growth restriction or who are small for gestational age (<10th percentile for weight) at birth.

Ages: 3 Days to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Ultrasound Transducer Compatibility | 1 year
  Successful acquisition and integration of a pediatric transducer with a footprint ≤ X cm² and focal depth ≤ Y mm (to be defined based on commercial availability and anatomical feasibility).
Hydrophone Sensitivity and Size | 1 year
  Selection and validation of a miniature hydrophone (e.g., diameter ≤ Z mm) with high sensitivity, characterized by its frequency response and minimum detectable pressure level.
Bandwidth Assessment | 1 year
  Measurement of hydrophone bandwidth (in MHz) as a primary indicator of sensitivity and signal capture quality.
System Performance Metrics | 1 year
  Quantitative assessment of signal-to-noise ratio (SNR) and resolution improvements compared to the previous setup using standard adult-sized components.
Feasibility in Preclinical Models | 1 year
  Demonstration of the optimized VAA system's ability to produce high-resolution, reproducible images in a neonatal bone phantom or relevant preclinical model.

SECONDARY OUTCOMES:
Quantitative Bone Health Index (BHI) | through the study completion, up to 3 years
  Derived from vibro-acoustic assessment (VAA) of the tibia in both term and preterm infants, BHI will be compared across age-adjusted groups to determine baseline differences between preterm and term infants.
VAA Sensitivity to Gestational Age | through the study completion, up to 3 years
  Correlation of VAA-derived parameters with gestational age at birth to assess the method's sensitivity in detecting bone development differences attributable to prematurity.
Longitudinal Changes in VAA Measurements | through the study completion, up to 3 years
  Assessment of VAA parameter changes over serial visits in preterm infants undergoing standard nutritional or medical interventions. Evaluates VAA's ability to detect improvements or deteriorations in bone status over time.
Comparison with Clinical Markers (if available) | through the study completion, up to 3 years
  Cross-validation of VAA findings with available clinical or biochemical markers of bone health (e.g., serum calcium, phosphate, ALP levels) to evaluate concurrent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT04752098/ICF_000.pdf